CLINICAL TRIAL: NCT02246075
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, 24-Week, Phase 2 Study of Two Doses of EVP-6124 Hydrochloride or Placebo in Subjects With Mild to Moderate Alzheimer's Disease Currently Receiving Memantine Medication With or Without Additional Acetylcholinesterase Inhibitor Co-Medication
Brief Title: Study of the Safety of Two Doses of Investigational Study Drug EVP-6124 in Subjects With Alzheimer's Disease Currently Receiving Memantine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Forum has decided not to proceed with this study at this time.
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-6124-027
Record Dates: First submitted 2014-09-17; First posted 2014-09-22 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-10

CONDITIONS: Alzheimer's Disease; Dementia; Cognition
Keywords: Alzheimer's disease; Cognition; Alpha-7 nAChR
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide; N-(7-chloro-N-quinuclidin-3-yl)benzo(b)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- EVP-6124, low dose (Experimental): Low dose, Tablet, Once Daily, Day 1 through Day 168
  Interventions: Drug: EVP-6124
- EVP-6124, high dose (Experimental): High dose, Tablet, Once Daily, Day 1 through Day 168
  Interventions: Drug: EVP-6124
- EVP-6124, Placebo (Placebo Comparator): Placebo, Tablet, Once Daily, Day 1 through Day 168
  Interventions: Drug: EVP-6124

INTERVENTIONS:
Drug: EVP-6124
  Other Names: encenicline

SUMMARY:
The purpose of this study is to evaluate the safety of 2 fixed doses of EVP-6124 hydrochloride (HCl) compared to placebo for 24 weeks in subjects with mild to moderate Alzheimer's disease who are concurrently receiving stable treatment with memantine and currently receiving stable treatment or previously treated with an acetylcholinesterase inhibitor.

ELIGIBILITY:
Inclusion Criteria:

* Ages ≥55 and ≤85 years
* Informed consent form (ICF) signed by the subject or legally acceptable representative before any study-specific procedures for the subject are performed and an ICF signed by the support person/caregiver before any study-specific procedures for the support person/caregiver are performed
* Clinical diagnosis of dementia due to possible or probable AD consistent with criteria established by a workgroup of the National Institute on Aging and the Alzheimer's Disease Association
* Magnetic resonance imaging (MRI) or computed tomography (CT) scan performed within 12 months before screening, with findings consistent with the diagnosis of dementia due to AD without any other clinically significant comorbid pathologies. If an MRI or CT scan is unavailable or occurred greater than 12 months before screening, this assessment should be completed and the findings confirmed before the subject enters the run-in period (Day -14) (copy of the report will be available at the study site)
* Mini-Mental State Examination (MMSE) score ≥12 and ≤26 at screening
* Modified Hachinski Ischemic Scale (mHIS) score ≤4 at screening
* Fertile, sexually active subjects (men and women) must use an effective method of contraception during the study. Female subjects and the female partner of male subjects must be surgically sterile (hysterectomy or bilateral tubal ligation), postmenopausal for at least 1-year, or willing to practice adequate methods of contraception if of childbearing potential (defined as consistent use of combined effective methods of contraception [including at least 1 barrier method])
* Reliable and capable support person/caregiver, who if not living in the same household, interacts with the subject regularly and will help facilitate clinic visits of the study subject
* Subject living at home, senior residential setting, or an institutional setting without the need for continuous (ie, 24-hour) nursing care
* General health status acceptable for participation in a 24-week study
* Fluency (oral and written) in the language in which the standardized tests will be administered
* Receiving a stable dose of memantine for at least 3 months (90 days) before screening and with continuous dosing for at least 3 months. Additional co-medication with an AChEI (donepezil in any dose form other than 23 mg once daily (QD), rivastigmine or galantamine) is allowed if stable for at least 3 months (90 days) before screening with total continuous exposure for at least 3 months.

Exclusion Criteria:

* Exposure to an experimental drug, experimental biologic or experimental medical device within 2 months (60 days) before screening
* Prior participation in an amyloid vaccination clinical study at any time in the past or completion of a passive amyloid vaccination study within 6 months before screening
* Inability to swallow a tablet
* In the judgment of the investigator, inability of the subject to complete a 24-week study
* Residence in a skilled nursing facility
* Inability to be ≥75% compliant with single-blind study drug
* Clinically significant (in the judgment of the investigator) abnormal serum electrolytes (sodium, potassium, magnesium) after repeat testing
* Clinically significant untreated hypothyroidism (if treated, thyroid-stimulating hormone level and thyroid supplementation dose must be stable for at least 6 months before screening)
* Insufficiently controlled diabetes mellitus (in the judgment of the investigator) or requiring insulin
* Renal insufficiency (serum creatinine >2.0 mg/dL)
* Malignant tumor within 3 years before screening (except squamous and basal cell carcinoma or cervical carcinoma in situ or localized prostate cancer)
* History of ischemic colitis or ischemic enterocolitis
* Unstable medical condition that is clinically significant in the judgment of the investigator
* Female subjects who are pregnant, nursing, or planning to become pregnant during the study
* Alanine transaminase (ALT) or aspartate transaminase (AST) >2.5 times the upper limit of normal
* History of myocardial infarction or unstable angina within 6 months before screening
* History of more than 1 myocardial infarction within 5 years before screening
* Clinically significant (in the judgment of the investigator) cardiac arrhythmia (including atrial fibrillation), cardiomyopathy, or cardiac conduction defect (subjects with a pacemaker are acceptable)
* Symptomatic hypotension, or uncontrolled hypertension (in the judgment of the investigator)
* Clinically significant abnormality on screening electrocardiogram (ECG), including but not necessarily limited to a confirmed QTc value ≥450 msec for males or ≥470 msec for females. In subjects with a QRS value >120msec, those with a QTc value <500 msec may be eligible following discussion with the Medical Monitor.
* Stroke within 18 months before screening, or history of a stroke concomitant with onset of dementia
* History of brain tumor, subdural hematoma, or other clinically significant (in the judgment of the investigator) space-occupying lesion on CT or MRI
* Head trauma with clinically significant (in the judgment of the investigator) loss of consciousness within 12 months before screening or concurrent with the onset of dementia
* Onset of dementia secondary (in the judgment of the investigator) to cardiac arrest, surgery with general anesthesia, or resuscitation
* Specific degenerative CNS disease diagnosis other than AD (eg, Huntington's disease, Creutzfeld-Jacob disease, Down's syndrome, Fronto-Temporal Dementia, Parkinson's disease)
* Wernicke's encephalopathy
* Active acute or chronic CNS infection
* Donepezil 23 mg QD currently or within 3 months prior to randomization
* Discontinued AChEI <30 days prior to randomization
* Antipsychotics; low doses (in the judgment of the investigator, except clozapine) are allowed only if given for sleep disturbances, agitation and/or aggression, and only if the subject has received a stable dose for at least 3 months before randomization
* Tricyclic antidepressants and monoamine oxidase inhibitors; all other antidepressants are allowed only if the subject has received a stable dose for at least 3 months before randomization
* Anxiolytics or sedative-hypnotics, including barbiturates (unless given in low doses for benign tremor); low doses of benzodiazepines and zolpidem (in the judgment of the investigator) are allowed only if given for insomnia/sleep disturbance, and only if the subject has received a stable dose for at least 3 months before randomization
* Peripherally acting drugs with effects on cholinergic transmission
* Immunosuppressants, including systemic corticosteroids, if taken in clinically immunosuppressive doses in the judgment of the investigator (Note: steroid use for allergy or other inflammation is permitted)
* Antiepileptic medications if taken for control of seizures
* Chronic intake of opioid-containing analgesics
* Sedating H1 antihistamines
* Nicotine therapy (all dosage forms including a patch), varenicline (Chantix), or similar therapeutic agent within 30 days before screening
* Clinically significant urine drug screen (UDS) or serum alcohol test result in the judgment of the investigator (including medical marijuana)

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Safety/Tolerability of EVP-6124 with concurrent memantine | Baseline to Day 168
  * Number of subjects with AEs
  * Percentage of subjects with AEs
  * Number of subjects with SAEs
  * Percentage of subjects with SAEs
  * Number of subjects who discontinue due to AEs
  * Percentage of subjects who discontinue due to AEs
  * Number of subject deaths
  * Percentage of subject deaths

SECONDARY OUTCOMES:
Change from Baseline in the Mini-Mental State Examination (MMSE) | Baseline to Day 168

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Delray Beach, Florida
  - Albuquerque, New Mexico